CLINICAL TRIAL: NCT06163586
Title: Effects of Neonatal Therapeutic Touch and Massage in Very Preterm and Extremely Preterm Neonates: A Randomized Controlled Trial
Brief Title: Massage Therapy in Premature Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Johana Diaz, Assistant professor of pediatrics, Division of neonatology, University of Maryland, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00098293
Record Dates: First submitted 2023-11-13; First posted 2023-12-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Neonatal Prematurity; Massage Therapy
Keywords: Prematurity; Massage therapy
MeSH Terms: conditions — Premature Birth | interventions — Massage

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessors evaluating neurodevelopmental outcomes will be masked from knowing which intervention was assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive structured neonatal touch or massage therapy from a certified NICU provider. Therapy will given 3 days a week for 5 to 15 minutes for a minimum of 4 weeks. We will also be collecting data to assess pain and stress responses during the period immediately before, during, and shortly after the therapy. This includes assessment of crying/irritability, behavior state, facial expression, extremities tone, and vital signs (heart rate, breathing rate, and oxygen levels).
  Interventions: Other: Neonatal Touch and Massage Therapy
- Control (No Intervention): This group will receive standard NICU care, no different than if they were not enrolled in the study.

INTERVENTIONS:
Other: Neonatal Touch and Massage Therapy — Structured touch and massage therapy performed by certified providers.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn about the effects of Neonatal Touch and Massage Therapy on premature babies.

The main questions it aims to answer are:

* Do babies who receive Neonatal Touch and Massage Therapy get discharged sooner from the NICU
* Does Neonatal Touch and Massage Therapy have a beneficial effect on weight gain, pain and stress responses, and neurodevelopmental outcomes.

Participants assigned to the treatment group will receive Neonatal Touch and Massage Therapy while admitted to the NICU. Researchers will compare their outcomes to a control group, receiving standard NICU care, to see if there are any differences in the length of hospital stay, weight gain, pain scores, neurodevelopmental outcomes, and incidence of other common conditions associated with prematurity.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of Neonatal Touch and Massage Therapy on premature infants in the NICU. Babies enrolled in this study will be randomly assigned to receive Neonatal Touch and Massage or standard NICU care. Babies in the therapy group will be given Neonatal Touch or Massage therapy by certified providers 3 days per week for 5 to 15 minutes. Therapy will be done for a minimum of 4 weeks. The investigators will assess pain and stress responses before and after treatment. The investigators will also review participant's medical records to collect information about weight gain, length of hospitalization, and general health status. After a participant is discharged home, information will be collected about participant's developmental assessments at regularly scheduled NICU follow-up clinic appointments. There are no significant risks with this therapy. Potential benefits of therapy include increased weight gain, shorter hospitalization, decreased pain and stress, and improved developmental outcomes. Information gained from this study could also help future babies.

ELIGIBILITY:
Inclusion Criteria:

* Infants born or admitted to University of Maryland NICU in the first 14 days of life
* Gestational age greater than 23 6/7 weeks and less than 32 weeks at birth
* Deemed medically stable by the medical care team

Exclusion Criteria:

* Life limiting conditions, including genetic syndromes
* Cyanotic heart disease
* Requiring major surgery or critically ill at time of intervention
* Osteopenia of prematurity with an existing fracture

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Length of stay | Day of birth to discharge home, up to 6 months
  Total length of hospitalization, from NICU admission to discharge home in days

SECONDARY OUTCOMES:
Weight gain | Through study intervention, an average of 4 weeks
  Assessment of daily weight in grams
Linear growth | Through study intervention, an average of 4 weeks
  Assessment of weekly length in centimeters
Head growth | Through study intervention, an average of 4 weeks
  Assessment of weekly head circumference in centimeters
Neurodevelopmental Outcomes | Within in 1 week of NICU discharge or transfer until up to 3 years of age
  Prior to NICU discharge or transfer each subject will undergo a Neonatal Neurobehavioral Scale (NNNS-II) assessment by a certified examiner. This is a comprehensive evaluation of neurological integrity and behavioral function including reflexes, motor development, and active and passive tone. NNNS profiles have been demonstrated to be predictive of short term cognitive, motor, and behavioral outcomes after NICU discharge. Standardized neurodevelopmental assessments will also be completed at regularly scheduled NICU follow-up clinic visits
Pain scores | 1 hour before intervention and up to 3 hours post-intervention
  Neonatal Pain, Agitation, and Sedation Scale (N-PASS) scores, a validated assessment tool using a combination of physiologic and behavioral indices, will documented before and after therapy to evaluate pain and stress responses. The scale has a minimum value of -10 and maximum value of +10, with a higher score indicating more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Johana Diaz, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Lago P, Garetti E, Merazzi D, Pieragostini L, Ancora G, Pirelli A, Bellieni CV; Pain Study Group of the Italian Society of Neonatology. Guidelines for procedural pain in the newborn. Acta Paediatr. 2009 Jun;98(6):932-9. doi: 10.1111/j.1651-2227.2009.01291.x. PMID 19484828
- [Background] Leslie Altimier, RN, MSN, DNPc, NEA-BC, Raylene M. Phillips, MD, MA, IBCLC, FAAP. The Neonatal Integrative Developmental Care Model: Seven Neuroprotective Core Measures for Family-Centered Developmental Care. Newborn & Infant Nursing Reviews 13 (2013) 9-22.
- [Background] Pickler RH, McGrath JM, Reyna BA, McCain N, Lewis M, Cone S, Wetzel P, Best A. A model of neurodevelopmental risk and protection for preterm infants. J Perinat Neonatal Nurs. 2010 Oct-Dec;24(4):356-65. doi: 10.1097/JPN.0b013e3181fb1e70. PMID 21045616
- [Background] Cruz MD, Fernandes AM, Oliveira CR. Epidemiology of painful procedures performed in neonates: A systematic review of observational studies. Eur J Pain. 2016 Apr;20(4):489-98. doi: 10.1002/ejp.757. Epub 2015 Jul 29. PMID 26223408
- [Result] Lai MM, D'Acunto G, Guzzetta A, Boyd RN, Rose SE, Fripp J, Finnigan S, Ngenda N, Love P, Whittingham K, Pannek K, Ware RS, Colditz PB. PREMM: preterm early massage by the mother: protocol of a randomised controlled trial of massage therapy in very preterm infants. BMC Pediatr. 2016 Aug 27;16(1):146. doi: 10.1186/s12887-016-0678-7. PMID 27568006
- [Result] Williams MD, Lascelles BDX. Early Neonatal Pain-A Review of Clinical and Experimental Implications on Painful Conditions Later in Life. Front Pediatr. 2020 Feb 7;8:30. doi: 10.3389/fped.2020.00030. eCollection 2020. PMID 32117835
- [Result] Badr LK, Abdallah B, Kahale L. A Meta-Analysis of Preterm Infant Massage: An Ancient Practice With Contemporary Applications. MCN Am J Matern Child Nurs. 2015 Nov-Dec;40(6):344-58. doi: 10.1097/NMC.0000000000000177. PMID 26302088
- [Result] Mrljak R, Arnsteg Danielsson A, Hedov G, Garmy P. Effects of Infant Massage: A Systematic Review. Int J Environ Res Public Health. 2022 May 24;19(11):6378. doi: 10.3390/ijerph19116378. PMID 35681968
- [Result] Niemi AK. Review of Randomized Controlled Trials of Massage in Preterm Infants. Children (Basel). 2017 Apr 3;4(4):21. doi: 10.3390/children4040021. PMID 28368368
- [Result] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Result] Alvarez MJ, Fernandez D, Gomez-Salgado J, Rodriguez-Gonzalez D, Roson M, Lapena S. The effects of massage therapy in hospitalized preterm neonates: A systematic review. Int J Nurs Stud. 2017 Apr;69:119-136. doi: 10.1016/j.ijnurstu.2017.02.009. Epub 2017 Feb 14. PMID 28235686
- [Result] McGowan EC, Hofheimer JA, O'Shea TM, Kilbride H, Carter BS, Check J, Helderman J, Neal CR, Pastyrnak S, Smith LM, Camerota M, Dansereau LM, Della Grotta SA, Lester BM. Analysis of Neonatal Neurobehavior and Developmental Outcomes Among Preterm Infants. JAMA Netw Open. 2022 Jul 1;5(7):e2222249. doi: 10.1001/jamanetworkopen.2022.22249. PMID 35849396
- [Result] Santos J, Pearce SE, Stroustrup A. Impact of hospital-based environmental exposures on neurodevelopmental outcomes of preterm infants. Curr Opin Pediatr. 2015 Apr;27(2):254-60. doi: 10.1097/MOP.0000000000000190. PMID 25635585
- [Result] Field T, Diego M, Hernandez-Reif M. Preterm infant massage therapy research: a review. Infant Behav Dev. 2010 Apr;33(2):115-24. doi: 10.1016/j.infbeh.2009.12.004. PMID 20137814
- [Result] Agarwal KN, Gupta A, Pushkarna R, Bhargava SK, Faridi MM, Prabhu MK. Effects of massage & use of oil on growth, blood flow & sleep pattern in infants. Indian J Med Res. 2000 Dec;112:212-7. PMID 11247199
- [Result] Arora J, Kumar A, Ramji S. Effect of oil massage on growth and neurobehavior in very low birth weight preterm neonates. Indian Pediatr. 2005 Nov;42(11):1092-100. PMID 16340050
- [Result] Fallah R, Akhavan Karbasi S, Golestan M, Fromandi M. Sunflower oil versus no oil moderate pressure massage leads to greater increases in weight in preterm neonates who are low birth weight. Early Hum Dev. 2013 Sep;89(9):769-72. doi: 10.1016/j.earlhumdev.2013.06.002. Epub 2013 Jul 5. PMID 23830725
- [Result] Saeadi R, Ghorbani Z, Shapouri Moghaddam A. The effect of massage with medium-chain triglyceride oil on weight gain in premature neonates. Acta Med Iran. 2015;53(2):134-8. PMID 25725185
- [Result] Wang L, He JL, Zhang XH. The efficacy of massage on preterm infants: a meta-analysis. Am J Perinatol. 2013 Oct;30(9):731-8. doi: 10.1055/s-0032-1332801. Epub 2013 Jan 15. PMID 23322391
- [Result] Vickers A, Ohlsson A, Lacy JB, Horsley A. Massage for promoting growth and development of preterm and/or low birth-weight infants. Cochrane Database Syst Rev. 2004;2004(2):CD000390. doi: 10.1002/14651858.CD000390.pub2. PMID 15106151
- [Result] Procianoy RS, Mendes EW, Silveira RC. Massage therapy improves neurodevelopment outcome at two years corrected age for very low birth weight infants. Early Hum Dev. 2010 Jan;86(1):7-11. doi: 10.1016/j.earlhumdev.2009.12.001. Epub 2009 Dec 22. PMID 20022717
- [Result] Fitri SYR, Nasution SK, Nurhidayah I, Maryam NNA. Massage therapy as a non-pharmacological analgesia for procedural pain in neonates: A scoping review. Complement Ther Med. 2021 Jun;59:102735. doi: 10.1016/j.ctim.2021.102735. Epub 2021 May 8. PMID 33974990
- [Result] Bernstein K, Karkhaneh M, Zorzela L, Jou H, Vohra S. Massage therapy for paediatric procedural pain: A rapid review. Paediatr Child Health. 2019 Nov 1;26(1):e57-e66. doi: 10.1093/pch/pxz133. eCollection 2021 Feb. PMID 33542780
- [Result] Hummel P, Puchalski M, Creech SD, Weiss MG. Clinical reliability and validity of the N-PASS: neonatal pain, agitation and sedation scale with prolonged pain. J Perinatol. 2008 Jan;28(1):55-60. doi: 10.1038/sj.jp.7211861. Epub 2007 Oct 25. PMID 18165830